CLINICAL TRIAL: NCT03226236
Title: Vaccination With Dendritic Cells Pulsed With Autologous Tumor Homogenate in Combination With HD-IL2 and Immunomodulating Radiotherapy in Metastatic RCC: a Phase II Trial (RENALVax-2)
Brief Title: Vaccination With Dendritic Cells Pulsed With Autologous Tumor Homogenate in Combination With HD-IL2 and Immunomodulating Radiotherapy in Metastatic RCC
Acronym: RENALVax-2
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No patients enrolled due to change in standard practice
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRST189.03; 2015-000556-14 (EudraCT Number)
Record Dates: First submitted 2016-09-28; First posted 2017-07-21 (Actual); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Carcinoma, Renal Cell; Vaccination; Secondary
Keywords: Carcinoma, Renal Cell; vaccination; dendritic cells; autologous tumor homogenate; High Dose -IL2; immunomodulating radiotherapy; secondary
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Metastasis | interventions — Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- study treatment (Experimental): boost radiotherapy (XRT) plus intradermal autologous dendritic cell vaccine loaded with autologous tumor homogenate (Autologous DC vaccine) plus High-Dose IL-2
  Interventions: Radiation: boost radiotherapy (XRT); Biological: Autologous DC vaccine; Drug: High-Dose IL-2

INTERVENTIONS:
Radiation: boost radiotherapy (XRT) — Three daily doses boost radiotherapy (XRT) at 6-12 Gy to at least 1, and up to a maximum of 5, metastatic fields, will be administrated on days -4 -3 -2 or -3 -2 -1 before the first and the third cycle of vaccine+IL-2
Biological: Autologous DC vaccine — The first dose (7 to 14 x 10_6 total dendritic cells) will be performed with freshly prepared vaccine, 9 days after leukapheresis; on day +1 starting from cycle 2 (3 weeks after the first cycle, on completion of QA assessments on the cryopreserved products), 5 additional doses will be administered every 3 weeks until maximum six vaccines.
Drug: High-Dose IL-2 — high dose IL-2: 18 MIU/m2/day in 500cc administered by continuous IV infusion for 72 hours starting day +2.

SUMMARY:
Single center, open-label Proof of Principle phase II trial to assess objective response (ORR).

Three daily doses boost radiotherapy (XRT) at 6-12 Gy to at least 1, and up to a maximum of 5, metastatic fields, will be administrated on days -4 -3 -2 or -3 -2 -1 before the first and the third cycle of vaccine+IL-2. The first day of administration of vaccine is day +1 and of IL-2 is day +2.

Treatment vaccine plus IL-2 (dose 18 MIU/m2/day in 500cc by continuous IV infusion for 72 hours) will be administered every 3 weeks up to 6 cycles.

Total duration of the trial: 36 months

* Enrolment period: 24 months
* Treatment: maximum of 6 cycles (5 months) per patient
* Follow-up every three months until patient died (follow-up until PD and only survival contacts and subsequent therapy for metastatic disease after PD).

DETAILED DESCRIPTION:
Vaccination with dendritic cells pulsed with autologous tumor homogenate in combination with HD-IL2 and immunomodulating radiotherapy in metastatic RCC: a phase II trial Proof of Principle phase II study Study Design Single center, open-label trial to assess response rate Study Duration Total duration: 36 months Enrollment: 24 months Treatment: 5 months per patient Follow-up every three months Primary objectives: Overall Response Rate (ORR) by irRC

Secondary end points:

1. Toxicity
2. Overall Survival
3. Duration of response
4. PFS
5. ORR by RECIST 1.1
6. Prognostic and predictive marker response
7. Immunological response Study Product, Dose, Route, Regimen and duration of administration Three daily doses boost radiotherapy (XRT) at 6-12 Gy to at least 1, and up to a maximum of 5, metastatic fields, will be administrated on days -4 -3 -2 or -3 -2 -1 before the first and the third cycle of vaccine+IL-2. The first day of administration of vaccine is day +1 and of IL-2 is day +2.

The intradermal autologous dendritic cell vaccine loaded with autologous tumor homogenate plus IL-2 (dose 18 MIU/m2/day in 500cc by continuous IV infusion for 72 hours) will be administered every 3 weeks up to 6 cycles.

Statistical Methodology

This is a Proof of Principle trial with a minimax two stage design:

• Step 1: 12 patients enrolled; A 5% response rate will preclude further study, whereas a 20% response rate will indicate that further study would be warranted.

Using alfa and beta errors of 0.10, if an objective response is observed in at least 1 of the 12 patients enrolled during the first stage the study will go on with a:

• Step 2: recruitment of an additional 25 patients The treatments will be considered active if an objective response is observed in 4 out of 37 patients treated.

The enrolment period will be 24 months. To ensure patients' safety, a continued safety evaluation by an independent DSMB will be performed and formal rules will be planned to continue or stop the recruitment; in particular, the enrollment will be interrupted when six patients completed at least one cycle of the combo treatment and they will be evaluated for safety: if grade ≥3 AEs (except for fever and rash that will be consider only for grade 4) in 2 (two) or more patients will be observed within 30 days after completion of the first dose of combo treatment, the study will be interrupted.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Written Informed Consent: patients must be willing and able to give written informed consent, that have to be given before starting of screening procedure.
2. Availability of autologous tumor tissue fulfilling acceptance criteria prescribed by the "Product Specification File".
3. Patients must have histologically or cytologically confirmed RCC (all histology types except for urothelial cancer);
4. Patients must have stage IV disease in progression after at least 1 TKI and/or antiangiogenetic and/or mTOR inhibitors therapy (patients must have finished prior treatments at least 4 weeks before the first IL2 dose)
5. Patients must have at least one measurable lesion, according to the irRC response criteria (see section 8 ), after asportation of tumor tissue for vaccine preparation. The tumor lesions that will be irradiated are excluded for response evaluation.
6. Life expectancy of greater than 3 months.
7. ECOG performance status 0-1
8. Patients must have organ and marrow function as defined below:

   * leukocytes >4000/µL
   * absolute neutrophil count >1,500/µL
   * platelets >100,000/µL
   * total bilirubin within normal institutional limits
   * AST(SGOT)/ALT(SGPT) <2.5 X institutional upper limit of normal
   * creatinine < 1.5 mg/dl
   * haemoglobin >8.0 gm/dl
   * hematocrit <30%
9. ECG and echocardiogram within normal institutional limits
10. Pulmonary function tests within normal institutional limits (to be performed only in patients with lung metastases or history of impaired lung function)
11. No contraindication for the use of vasopressor agents
12. Negative screening tests for HIV, HBV HCV and syphilis not older than 30 days before performing any of the GMP-regulated activities required (leukapheresis, collection of tumor biopsies to be used for tumor homogenate preparation);
13. Men and women aged > 18 years.
14. Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up 8 weeks after the study, in order to minimize the risk of pregnancy;
15. Patients must have normal organ and marrow function according to clinical practice.

Exclusion Criteria:

1. Patients who have positive tests to HCV, HBV, HIV, or syphilis (specific blood testing must be performed within 30 days before any GMP-regulated activity (leukapheresis and collection of tumor biopsies to be used for tumor homogenate preparation).
2. Patients who did not have prior lines of systemic therapy for advanced disease.
3. Participation in another clinical trial with any investigational agents within 30 days prior to study screening.
4. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements (on physician's judgment).
5. Other known malignant neoplastic diseases in the patient's medical history with a disease-free interval of less than 3 years (except for previously treated basal cell carcinoma and in situ carcinoma of the uterine cervix);
6. Patients who have had chemotherapy or radiotherapy or immunotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
7. Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
8. History of allergic reactions attributed to compounds of similar chemical or biologic composition to IL-2 or other agents used in the study.
9. Any autoimmune disease which could be exacerbated by IL-2
10. A medical illness requiring chronic treatments with corticosteroids or other immunosuppressive agents
11. A history of significant cardiovascular disease, including myocardial infarction, congestive heart failure, primary cardiac arrhythmias, angina pectoris or cerebrovascular accident
12. HIV-positivity, whether or not symptomatic
13. Any contraindication to undergo leukapheresis as evaluated by transfusionist (e.g. severe anemia, piastrinopenia, oral anticoagulant therapy) or to undergo surgery.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) by Immune related Response Criteria( irRC) | up to 24 months
  The analysis will be performed on an intention to treat population, i.e. all patients having received at least 2 cycles of therapy.

SECONDARY OUTCOMES:
Overall survival (OS) | up to 24 months
  measured from the date of registration until the date of death from any cause or the last date the patient was known to be alive and will be estimated with Kaplan-Meier method and the log rank test
Duration of response | up to 24 months
  time calculated from documentation of tumor response to disease progression
Progression free survival | up to 24 months
  measured from registration until disease progression or death
Immunologic efficacy | up to 24 months
  Immunologic efficacy will be measured by best DTH score (reactivity to homogenate or KLH) obtained after at least 4 vaccine doses, alone or combined with IFN-g ELISPOT analysis of tumor antigen-specific circulating effectors obtained after a minimum of 4 vaccine doses, both compared with prevaccine samples
Adverse events evaluation | up to 24 months
  Number of patients with treatment related Adverse events (AE) will be evaluated by CTCAE v 4.03 criteria The percentage of patients reporting an AE up to 30 days after HD-IL-2 treatment will be tabulated with 95% confidence intervals, by type of AE. The overall rate of grade 3-4 related AE will be computed

CONTACTS AND LOCATIONS:
Overall Officials: Laura Ridolfi, MD, Principal Investigator — UO Immunoterapia e Laboratorio TCS, Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST) S.r.l IRCCS
Locations (1):
- UO Immunoterapia e Laboratorio TCS, IRCCS IRST, Meldola (FC), FC, Italy

IPD SHARING:
Plan to Share IPD: Undecided